CLINICAL TRIAL: NCT06620575
Title: Evaluation of Predictive Factors for Recurrence of Persistent Atrial Fibrillation After Ablation
Acronym: FAIR
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-12-033
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Persistent atrial fibrillation ablation

SUMMARY:
This is a single-center, retrospective, observational study based on data extracted from the medical records of patients who underwent a procedure for persistent atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older, who has been informed about the research
* Patient who underwent a procedure for persistent atrial fibrillation ablation at Clairval Hospital since January 2014
* Patient for whom data regarding the ablation procedure are available

Exclusion criteria:

* Patient under legal protection, guardianship, or conservatorship
* Patient who has expressed opposition to the use of their medical data (by completing and returning the opt-out form provided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who underwent a procedure for persistent atrial fibrillation ablation at Clairval Hospital since January 2014
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Recurrence of persistent atrial fibrillation | Month 12
  The main objective of the study is to assess to what extent patient characteristics and conditions during the atrial fibrillation ablation procedure can identify predictive factors for recurrence.
  Recurrence (Yes/No) is the outcome variable to be explained.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Clairval, Marseille, France

IPD SHARING:
Plan to Share IPD: No